CLINICAL TRIAL: NCT04865978
Title: Evaluation of the Hemocompatibility of the Direct Oral Anti-Coagulant Apixaban in Left Ventricular Assist Devices
Acronym: DOAC LVAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palak Shah (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, Palak Shah, Medical Director, Mechanical Circulatory Support, Inova Health Care Services
Organization: Inova Health Care Services (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U21-06-4470
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
Keywords: ventricular assist device; LVAD; anticoagulation; apixaban; warfarin
MeSH Terms: conditions — Heart Failure | interventions — apixaban; Warfarin

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, randomized, 1:1 intervention arm versus control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Apixaban (Experimental): LVAD patients randomized to the experimental arm will be prescribed apixaban 5 mg twice daily.
  Interventions: Drug: Apixaban; Device: LVAD implant
- Warfarin (Active Comparator): LVAD patients randomized to the control arm will be prescribed warfarin which will be dosed to achieve an INR goal of 2-2.5
  Interventions: Drug: Warfarin; Device: LVAD implant

INTERVENTIONS:
Drug: Apixaban — Patients randomized to apixaban will be started on a dose of 5 mg BID.
  Arms: Apixaban
Drug: Warfarin — Patients randomized to warfarin will be started on a dose per institutional protocol and titrated to an INR goal of 2.0 - 2.5.
  Arms: Warfarin
Device: LVAD implant — Subjects will undergo HeartMate 3 LVAD implant prior to randomization

SUMMARY:
Prospective, randomized, controlled, open label, trial of LVAD patients with 1:1 randomization to either apixaban or warfarin.

DETAILED DESCRIPTION:
This pilot study will be a prospective, randomized, controlled, open label, trial of HeartMate 3 (HM3) LVAD patients with 1:1 randomization to either apixaban or warfarin. All patients will be treated with aspirin 81 mg daily as per the LVAD manufacturer instructions for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

1. Patients implanted with a HeartMate 3 LVAD
2. Age 18 or greater and able to provide written informed consent
3. Females of childbearing age must agree to adequate contraception

Exclusion Criteria:

1. History of post-LVAD device thrombosis, stroke, or gastrointestinal bleeding
2. Patients who are bridge to transplant and a current UNOS status 1-3
3. Ongoing inotrope therapy after LVAD (e.g., milrinone, dobutamine, epinephrine)
4. Permanent right ventricular assist device at the time of LVAD implant
5. Patients with a mechanical heart valve
6. Patients with end-stage renal disease on dialysis
7. Pregnant patients
8. Known history of ischemic stroke, intracranial bleed, or neurosurgery within 3 months
9. Known history of intracerebral arteriovenous malformation, cerebral aneurysm or mass lesions of the central nervous system.
10. Recent (<48 hours) or planned spinal or epidural anesthesia or puncture
11. Prior history of known thrombophilia (e.g., factor V Leiden, prothrombin gene mutation, protein C or S deficiency, antithrombin 3 deficiency, hyperhomocysteinemia, antiphospholipid antibody syndrome) or indication for higher INR goal (>2.5) with warfarin.
12. Thrombolysis within the previous 7 days
13. Patients with an allergy or contraindication to aspirin, warfarin, or apixaban
14. Patients on antiplatelet therapy other than aspirin (e.g., clopidogrel, prasugrel, ticagrelor, dipyridamole, or pentoxifylline)
15. Patients on combined P-glycoprotein and strong CPY3A4 inhibitors or inducers (e.g., fluconazole, posaconazole, rifampin)
16. Known bleeding within the last 30 days requiring emergency room presentation or hospitalization
17. Known history of an inherited bleeding disorder (e.g., hemophilia, von Willebrand disease)
18. Patients with active bleeding or a hemoglobin < 8.0 g/dl
19. Total bilirubin > 2.0 mg/dl, shock liver, hepatic encephalopathy, or biopsy proven liver cirrhosis
20. INR > 2.0 not due to anticoagulation therapy
21. Platelet count <100,000 cells/mm3

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Palak Shah, MD, MS, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimond M, Looby M, Shah B, Sinha SS, Isseh I, Rollins AT, Abdul-Aziz AA, Kennedy J, Tang DG, Klein KM, Casselman S, Vermeulen C, Sheaffer W, Snipes M, O'connor CM, Shah P. Design and Rationale for the Direct Oral Anticoagulant Apixaban in Left Ventricular Assist Devices (DOAC LVAD) Study. J Card Fail. 2024 Jun;30(6):819-828. doi: 10.1016/j.cardfail.2023.10.473. Epub 2023 Nov 11. PMID 37956897
- [Result] Shah P, Looby M, Dimond M, Bagchi P, Shah B, Isseh I, Rollins AT, Abdul-Aziz AA, Kennedy J, Tang DG, Klein KM, Casselman S, Vermeulen C, Sheaffer W, Snipes M, Sinha SS, O'Connor CM. Evaluation of the Hemocompatibility of the Direct Oral Anticoagulant Apixaban in Left Ventricular Assist Devices: The DOAC LVAD Study. JACC Heart Fail. 2024 Sep;12(9):1540-1549. doi: 10.1016/j.jchf.2024.04.013. Epub 2024 May 7. PMID 38795110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 16 | 14
Completed | 15 | 14
Not Completed | 1 | 0
Not completed — One patient did not complete the study due to infection and device explant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [49 to 75] | 56 [52 to 64] | 60 [52 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnic Group: White | 11 | 2 | 13
  Race or Ethnic Group: Black | 3 | 11 | 14
  Race or Ethnic Group: Asian | 1 | 1 | 2
  Race or Ethnic Group: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Death or Hemocompatibility Related Adverse Events (Stroke, Device Thrombosis, Bleeding, Aortic Root Thrombus, and Arterial Non-CNS Thromboembolism)
Description: Freedom from death or hemocompatibility related adverse events (composite of stroke, device thrombosis, bleeding, aortic root thrombus, and arterial non-CNS thromboembolism)
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 12

2. Secondary Outcome: Survival Free of Any Stroke
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

3. Secondary Outcome: Survival Free of Ischemic Stroke
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

4. Secondary Outcome: Survival Free of Hemorrhagic Stroke
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

5. Secondary Outcome: Survival Free of Device Thrombosis
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

6. Secondary Outcome: Survival Free of Gastrointestinal Bleeding
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 12

7. Secondary Outcome: Survival Free of Major Non-gastrointestinal Bleeding
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

8. Secondary Outcome: All-cause Mortality
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

9. Secondary Outcome: Cardiovascular Mortality
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

10. Secondary Outcome: Survival Free of Aortic Root Thrombus
Description: Compared between each study arm
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

11. Other Pre Specified Outcome: Freedom From Death or Hemocompatibility Related Adverse Events Evaluated in Subgroups of Patients Within 3 Months of Implant Versus Greater Than 3 Months From LVAD Implant
Description: Freedom From Death or Hemocompatibility Related Adverse Events (composite of Stroke, Device Thrombosis, Bleeding, Aortic Root Thrombus, and Arterial Non-CNS Thromboembolism) evaluated in subgroups of patients within 3 months of implant versus greater than 3 months from LVAD implant
Time Frame: From enrollment to end of treatment at 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Apixaban, Less Than 3 Months Since LVAD Implantation; Apixaban, 3 or More Months Since LVAD Implantation: LVAD patients randomized to the experimental arm will be prescribed apixaban 5 mg twice daily.
  Apixaban: Patients randomized to apixaban will be started on a dose of 5 mg BID.
  LVAD implant: Subjects will undergo HeartMate 3 LVAD implant prior to randomization
- Warfarin, Less Than 3 Months Since LVAD Implantation; Warfarin, 3 or More Months Since LVAD Implantation: Patients randomized to warfarin will be started on a dose per institutional protocol and titrated to an INR goal of 2.0 - 2.5.
  Subjects will undergo HeartMate 3 LVAD implant prior to randomization
Arm/Group | Apixaban, Less Than 3 Months Since LVAD Implantation | Apixaban, 3 or More Months Since LVAD Implantation | Warfarin, Less Than 3 Months Since LVAD Implantation | Warfarin, 3 or More Months Since LVAD Implantation
Number analyzed (Participants) | 8 | 8 | 6 | 8
Participants | 8 | 8 | 5 | 7

ADVERSE EVENTS:
Time Frame: From enrollment to final safety visit at 28 weeks
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 7/16 | 8/14
Other Adverse Events (participants affected / at risk) | 14/16 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=16) | Warfarin (N=14)
Serious AE Infection (Infections and infestations) | 4 (5) | 3 (3) — Infection requiring hospitalization
Serious AE Cardiac (Cardiac disorders) | 2 (2) | 1 (1) — Hospitalization for heart failure
Serious AE Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 3 (4) — Gastrointestinal bleeding, serious
Serious AE Other (General disorders) | 1 (1) | 4 (4) — Other serious adverse events included in the warfarin group include (1 each): diabetic ketoacidosis, arrhythmia, severed driveline, RV thrombus; Other serious adverse events included in the apixaban group includes (1 each): hypertensive urgency
Serious AE Device Related (Surgical and medical procedures) | 1 (1) | 0 (0) — Device explant
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=16) | Warfarin (N=14)
AE Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1) | 0 (0)
AE Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
AE Hematologic (Blood and lymphatic system disorders) | 10 (17) | 3 (3)
AE Infection (Infections and infestations) | 6 (7) | 4 (4)
AE Cardiac (Cardiac disorders) | 9 (9) | 8 (9)
AE Neurologic (Nervous system disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT04865978/Prot_SAP_000.pdf